CLINICAL TRIAL: NCT02909114
Title: Phase II Study of Stereotactic Body Radiotherapy for Oligometastases From Colorectal Cancer
Brief Title: Stereotactic Body Radiotherapy for Oligometastases From Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jing Jin, M.D. (Unknown)
Responsible Party: Sponsor-Investigator, Jing Jin, M.D., Medical Doctor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-096
Record Dates: First submitted 2016-09-12; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Colorectal Cancer
Keywords: stereotactic boday radiotherapy, oligometastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental group (Experimental): SBRT for oligometastatases from colorectal cancer objectives
  Interventions: Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — All patients will undergo planning CT simulation. 4-dimensional CT will be used for tumors in the lungs or liver. For all lesions, the gross tumor volume (GTV) will be defined as the visible tumor on CT and/or MRI imaging +/- PET. A Planning Target Volume (PTV) margin of 3-5 mm will be added depending on site of disease, immobilization, and institutional set-up accuracy.
  The prescirbe dosage was as following: Lung lesion DT50-60 Gy/5 fractions; liver 50-60Gy/5-8 fractions; brain DT 40Gy/4-5fractions. All will be treated with SBRT

SUMMARY:
Single arms prospective phase II study of SBRT for oligometastatases from colorectal cancer

DETAILED DESCRIPTION:
Single arms prospective phase II study of SBRT for oligometastatases from colorectal cancer, the primary concerns are treatment efficacy and toxicities.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years
* Eastern Cooperative Oncology Group (ECOG) performance score ≤ 1
* Diagnosis by pathological examination
* Primary lesion is under control by surgery
* Adequate blood counts:

  * White blood cell count ≥3.5 x 109/L
  * Haemoglobin levels ≥100g/L
  * Platelet count ≥100 x 109/L
  * Creatinine levels ≤1.0× upper normal limit (UNL)
  * Urea nitrogen levels ≤1.0× upper normal limit (UNL)
  * Alanine aminotransferase (ALT) ≤1.5× upper normal limit (UNL)
  * Aspartate aminotransferase (AST) ≤1.5× upper normal limit (UNL)
  * Alkaline phosphatase (ALP) ≤1.5× upper normal limit (UNL)
  * Total bilirubin (TBIL) ≤1.5× upper normal limit (UNL)

Exclusion Criteria:

* Primary lesion is not under control
* Pancreatic carcinoma
* Oligometastases could not be located
* Pregnancy or breast feeding
* Symptoms or history of peripheral neuropathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
local control assessed by RECIST | 3 years

SECONDARY OUTCOMES:
>= Grade 3 treatment-related adverse events as assessed by CTCAE v4.0 | from radiotherapy start to complete treatment 90 days
overall survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Acadamy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes